CLINICAL TRIAL: NCT06282679
Title: Clinical Observation of Intradermal Injections With Botulinum Toxin A in the Treatment of Rosacea Erythema Telangiectasia
Brief Title: Clinical Observation of Botulinum Toxin A Treatment in the Treatment of Rosacea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, dai jie, Nanjing First Hospital, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20220701-03
Record Dates: First submitted 2023-04-05; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Rosacea; Botulinum Toxin
MeSH Terms: conditions — Rosacea | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- left cheek and right cheek (Experimental): First, apply an appropriate amount of lidocaine cream to your face and wait (30-45 minutes) for the anesthetic to take effect;
  Second step, after cleaning, mark the injection site on your face, about 25-30 points on one cheek, 1 cm apart, using a randomized half face control trial, Use of botulinum toxin type A for injection (Botox) (Allergan Pharmaceticals Ireland Limited, Import Drug Registration No. : S20171003), 0.5U botulinum toxin type A (Botox) was injected per point on one cheek and 1U on the other. The total amount of botulinum toxin type A was between 15 and 30U on each side.
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection [Botox] — you are asked to return to the hospital for follow-up at weeks 2, 4, 8, and 12
  Other Names: follow

SUMMARY:
the goal of this study is to study the clinical efficacy and safety of botox in the treatment of rosacea.

DETAILED DESCRIPTION:
The main objective is to collect patients and then use different injection volumes of botulinum toxin intradermal injection for the treatment of rosacea erythema telangiectasia, and then to evaluate the clinical efficacy and safety of the treatment.

ELIGIBILITY:
Inclusion Criteria

* Meeting the diagnostic criteria of mild to moderate erythema telangiectasis rosette acne;
* more than 18 years old;
* to obey the rules of the treatment in the study, and can be followed up for 12 weeks;
* informed consent;

Exclusion Criteria:

* Had received facial cosmetic surgery or botulinum toxin treatment within 6 months before this treatment;
* due to systemic diseases such as autoimmune diseases or menopause facial flush;
* had allergies botulinum toxin;
* pregnant or breastfeeding;
* other facial skin or oral disease therapy, including research before 4 weeks rose acne accept other treatment;
* With basic neuromuscular diseases (such as myasthenia gravis, amyotrophic lateral sclerosis, etc.);
* All landowners 4 weeks before the study whether any oral aminoglycoside drugs, benzodiazepines drugs or muscle relaxants; .Was removed during treatment observation data is not complete, incomplete treatment and patients can't take medication as prescribed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
CEA score | 2.4,8,12 weeks
  Clinical erythema score (CEA) was divided into no, mild, moderate and severe according to the severity of rosacea, corresponding to 0,1,2,3, respectively

SECONDARY OUTCOMES:
GAIS score | 2.4,8,12 weeks
  he Global Aesthetic Improvement Scale (GAIS) score was assessed by the treating physician on the patient's improvement and was divided into four levels: very improved corresponding, substantial improvement, improvement, no change; Corresponding to the best beauty results, significantly improved but not the best, significantly improved, no change

OTHER OUTCOMES:
VISIA red zone score | 2.4,8,12 weeks
  VISIA Red zone score The patient's face was photographed by VISIA analyzer and corresponding indicators such as feature index and percentage were recorded
Dermatology Quality of Life Score (DLQI) | 2.4,8,12 weeks
  The Dermatology Life Quality Score (DLQI) is scored by answering multiple questions in which patients self-rate the impact of their current illness on their lives over a period of one week. The answer is divided into four levels, very serious 3 points, severe 2 points, a little 1 point, no 0 points;

CONTACTS AND LOCATIONS:
Overall Officials: Jie DAI, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jie Dai, Nanjing, Jiangsu, China

REFERENCES:
- [Result] van Zuuren EJ. Rosacea. N Engl J Med. 2017 Nov 2;377(18):1754-1764. doi: 10.1056/NEJMcp1506630. No abstract available. PMID 29091565
- [Result] Marson JW, Baldwin HE. Rosacea: a wholistic review and update from pathogenesis to diagnosis and therapy. Int J Dermatol. 2020 Jun;59(6):e175-e182. doi: 10.1111/ijd.14757. Epub 2019 Dec 27. PMID 31880327
- [Result] Moustafa F, Lewallen RS, Feldman SR. The psychological impact of rosacea and the influence of current management options. J Am Acad Dermatol. 2014 Nov;71(5):973-80. doi: 10.1016/j.jaad.2014.05.036. Epub 2014 Jul 1. PMID 24993600
- [Result] Gallo RL, Granstein RD, Kang S, Mannis M, Steinhoff M, Tan J, Thiboutot D. Standard classification and pathophysiology of rosacea: The 2017 update by the National Rosacea Society Expert Committee. J Am Acad Dermatol. 2018 Jan;78(1):148-155. doi: 10.1016/j.jaad.2017.08.037. Epub 2017 Oct 28. PMID 29089180
- [Result] Bloom BS, Payongayong L, Mourin A, Goldberg DJ. Impact of intradermal abobotulinumtoxinA on facial erythema of rosacea. Dermatol Surg. 2015 Jan;41 Suppl 1:S9-16. doi: 10.1097/DSS.0000000000000277. PMID 25548852
- [Result] Schwab VD, Sulk M, Seeliger S, Nowak P, Aubert J, Mess C, Rivier M, Carlavan I, Rossio P, Metze D, Buddenkotte J, Cevikbas F, Voegel JJ, Steinhoff M. Neurovascular and neuroimmune aspects in the pathophysiology of rosacea. J Investig Dermatol Symp Proc. 2011 Dec;15(1):53-62. doi: 10.1038/jidsymp.2011.6. PMID 22076328
- [Result] Holowatz LA, Thompson CS, Minson CT, Kenney WL. Mechanisms of acetylcholine-mediated vasodilatation in young and aged human skin. J Physiol. 2005 Mar 15;563(Pt 3):965-73. doi: 10.1113/jphysiol.2004.080952. Epub 2005 Jan 20. PMID 15661816
- [Result] Choi JE, Werbel T, Wang Z, Wu CC, Yaksh TL, Di Nardo A. Botulinum toxin blocks mast cells and prevents rosacea like inflammation. J Dermatol Sci. 2019 Jan;93(1):58-64. doi: 10.1016/j.jdermsci.2018.12.004. Epub 2018 Dec 28. PMID 30658871
- [Result] Huang W, Foster JA, Rogachefsky AS. Pharmacology of botulinum toxin. J Am Acad Dermatol. 2000 Aug;43(2 Pt 1):249-59. doi: 10.1067/mjd.2000.105567. PMID 10906647
- [Result] Kim MJ, Kim JH, Cheon HI, Hur MS, Han SH, Lee YW, Choe YB, Ahn KJ. Assessment of Skin Physiology Change and Safety After Intradermal Injections With Botulinum Toxin: A Randomized, Double-Blind, Placebo-Controlled, Split-Face Pilot Study in Rosacea Patients With Facial Erythema. Dermatol Surg. 2019 Sep;45(9):1155-1162. doi: 10.1097/DSS.0000000000001819. PMID 30730346
- [Result] Dayan SH, Ashourian N, Cho K. A Pilot, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of IncobotulinumtoxinA Injections in the Treatment of Rosacea. J Drugs Dermatol. 2017 Jun 1;16(6):549-554. PMID 28686772
- [Result] Eshghi G, Khezrian L, Alirezaei P. Botulinum Toxin A in Treatment of Facial Flushing. Acta Med Iran. 2016 Jul;54(7):454-7. PMID 27424017
- [Result] Serarslan G, Makbule Kaya O, Dirican E. Scale and Pustule on Dermoscopy of Rosacea: A Diagnostic Clue for Demodex Species. Dermatol Pract Concept. 2021 Jan 29;11(1):e2021139. doi: 10.5826/dpc.1101a139. eCollection 2021 Jan. PMID 33614217
- [Result] Sharma A, Kroumpouzos G, Kassir M, Galadari H, Goren A, Grabbe S, Goldust M. Rosacea management: A comprehensive review. J Cosmet Dermatol. 2022 May;21(5):1895-1904. doi: 10.1111/jocd.14816. Epub 2022 Feb 14. PMID 35104917